CLINICAL TRIAL: NCT00372021
Title: Neurotomy of Optic Nerve in Non-Arthritic Anterior Ischemic Optic Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8136
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2002-11

CONDITIONS: Non Arthritic Anterior Ischemic Optic Neuropathy
Keywords: non arthritic ischemic optic neuropathy; anterior ischemic optic neuropathy; Optic nerve Neurotomy
MeSH Terms: conditions — Optic Neuropathy, Ischemic

INTERVENTIONS:
Procedure: optic nerve neurotomy

SUMMARY:
Non-arthritic anterior ischemic optic neuropathy is the most common cause of sudden visual loss due to optic nerve involvement in patients above 50 years old. As this problem can be considered as a sclera out let syndrome an there is no effective and successful treatment for it, we decided to do a neurotomy procedure and relax the involved optic nerve in order to achieve acceptable treating outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-arthritic anterior ischemic optic nerve

Exclusion Criteria:

* Visual acuity more than 20/200
* Other intra occular operations
* Passing more than 4 weeks of the problem
* Arthritic anterior ischemic optic nerve
* Age under 50 years
* Consumption of previous pharmaceutical treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-01

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Soheilian, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran